CLINICAL TRIAL: NCT01270672
Title: Effects of Carvedilol on the Cardiovascular and Subjective Response to MDMA (3,4-Methylenedioxymethamphetamine, "Ecstasy")
Brief Title: Pharmacological Interaction Between Carvedilol and Methylenedioxymethamphetamine (MDMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 218/10
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Mood Disorder; Substance-Related Disorders; Amphetamine-Related Disorders
Keywords: MDMA; carvedilol; norepinephrine; alpha - beta receptor; Ecstasy; stimulant
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carvedilol, MDMA, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: carvedilol; Drug: placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 125 mg per os, single dose
  Other Names: MDMA; Ecstasy; Adam
Drug: carvedilol — 50 mg per os, single dose
Drug: placebo — capsules identical to MDMA or carvedilol

SUMMARY:
The purpose of this study is to determinate the effect of a pre-treatment with carvedilol, a alpha- and beta-adrenergic receptor blocker, on the pharmacodynamics and pharmacokinetics of 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy"). The investigators hypothesize that carvedilol will attenuate the cardiovascular and subjective response to MDMA.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), dopamine, and norepinephrine (NE). NE release is thought to mediate the cardiovascular effects of MDMA and may also contribute to its psychostimulant effects. However, the functional role of adrenergic postsynaptic receptors in the cardiovascular and subjective effects of MDMA in humans is largely unclear. To determine the role of alpha- and beta adrenergic receptors in the response to MDMA in humans the investigators test the effects of the alpha- and beta-receptor blocker carvedilol on the physiological and subjective effects of MDMA. The investigators use a randomized double-blind placebo-controlled cross-over design with four experimental sessions. Carvedilol or placebo will be administered 1 h before MDMA or placebo to 16 healthy volunteers. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics. The primary hypothesis is that carvedilol will significantly reduce the blood pressure response to MDMA.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except Tetrahydrocannabinol-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Effect of carvedilol on the blood pressure response to MDMA | 24 h

SECONDARY OUTCOMES:
Effect of carvedilol on the subjective response to MDMA | 24 h
Effect of carvedilol on neuroendocrine effects of MDMA | 7 h
Effect of carvedilol on pharmacokinetics of MDMA | 7 h

OTHER OUTCOMES:
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — Department of Internal Medicine, Division of Pharmacology & Toxicology, University Hospital Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Liechti ME. Effects of MDMA alone and after pretreatment with reboxetine, duloxetine, clonidine, carvedilol, and doxazosin on pupillary light reflex. Psychopharmacology (Berl). 2012 Dec;224(3):363-76. doi: 10.1007/s00213-012-2761-6. Epub 2012 Jun 15. PMID 22700038